CLINICAL TRIAL: NCT04738331
Title: Analysing the French COVID-19 Epidemic Using a National SARS-CoV-2 RT-PCR Database : CovPCR
Brief Title: Analysing the French COVID-19 Epidemic Using a National SARS-CoV-2 RT-PCR Database
Acronym: CovPCR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0051
Record Dates: First submitted 2021-02-02; First posted 2021-02-04 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Covid-19; SARS-CoV Infection
Keywords: SARS-Cov2 infection; Tested for SARS-Cov2 infection with RT-PCR test; CT; epidemiology; reproduction number
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Analysing ths spread of COVID-19 epidemics in a timely manner is key to implementing public health control strategies. The investigators propose to analyse a large set of laboratory SARS-CoV-2 RT-PCR data to explore potential links between Ct values and epidemic parameters.

ELIGIBILITY:
Inclusion criteria:

- A SARS-Cov2 RT-PCR result with a known sampling date

Exclusion criteria:

- Patient refusing to participate in research

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: French population with a RT-PCR test for SARS-Cov2 infection
Sampling Method: Non-Probability Sample
Enrollment: 10000000 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-05-20 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Detecting co-factors associated with Ct values | 1 day
  Detecting co-factors associated with Ct values

SECONDARY OUTCOMES:
Detecting associations with epidemic spread | 1 day
  Detecting associations with epidemic spread

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Foulongne, PhD, Study Director — UH MONTPELLIER
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC